CLINICAL TRIAL: NCT04104672
Title: A Phase 1 Study to Evaluate the Safety and Tolerability of AB680 Combination Therapy in Participants With Gastrointestinal Malignancies
Brief Title: A Study to Evaluate the Safety and Tolerability of AB680 in Participants With Gastrointestinal Malignancies
Acronym: ARC-8
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARC-8 (AB680CSP0002)
Record Dates: First submitted 2019-09-23; First posted 2019-09-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-05

CONDITIONS: Advanced Pancreatic Cancer
Keywords: AB680; Zimberelimab; Pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — quemliclustat; zimberelimab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Intervention Model Description: 3+3 Dose escalation design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Dose Escalation (Experimental): Dose escalation is a 3+3 design, including a Dose Limiting Toxicity (DLT) evaluation period. The dose expansion dose level will be determined in this part with escalating doses of AB680 in combination with zimberelimab at the recommended phase 2 dose (RP2D) and the standard nab-paclitaxel and gemcitabine chemotherapy regimen in participants with advanced pancreatic cancer.
  Interventions: Drug: AB680; Drug: Zimberelimab; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Dose Expansion (AB680+zimberelimab+ NP/Gem): Cohort A (front-line/1L) (Experimental): Participants with advanced pancreatic cancer, naïve to any prior treatment will receive AB680 (at the RP2D identified during dose escalation) combined with zimberelimab and the standard nab-paclitaxel (NP) and gemcitabine (Gem) (NP/Gem) chemotherapy regimen
  Interventions: Drug: AB680; Drug: Zimberelimab; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Dose Expansion (AB680+zimberelimab+NP/Gem):Cohort A1 (front-line/1L) (Experimental): Participants with advanced pancreatic cancer, naïve to any prior treatment will receive AB680 (at the RP2D identified during dose escalation) combined with zimberelimab and the standard nab-paclitaxel (NP) and gemcitabine (Gem) (NP/Gem) chemotherapy regimen
  Interventions: Drug: AB680; Drug: Zimberelimab; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Dose Expansion (AB680 + NP/Gem): Cohort A2 (front-line/1L) (Experimental): Participants with advanced pancreatic cancer who are naïve to any prior treatment will receive AB680 (at the RP2D identified during dose escalation) and the standard NP/Gem chemotherapy regimen.
  Interventions: Drug: AB680; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Dose Expansion (AB680 + zimberelimab + NP/Gem): Cohort B (second-line/2L) (Experimental): Participants with advance pancreatic cancer who have received 1 prior line of treatment will receive AB680 (at the RP2D identified during dose escalation) combined with zimberelimab and NP-Gem chemotherapy regimen.
  Interventions: Drug: AB680; Drug: Zimberelimab; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Dose Expansion (AB680 + zimberelimab + NP/Gem): Cohort C (front-line/1L) (Experimental): Participants with advanced pancreatic cancer naïve to any prior treatment will receive AB680 combined with zimberelimab and NP-Gem chemotherapy regimen.
  Interventions: Drug: AB680; Drug: Zimberelimab; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Dose Expansion (AB680 + NP/Gem): Cohort D (front-line/1L) (Experimental): Participants with advanced pancreatic cancer naïve to any prior treatment will receive AB680 combined with NP-Gem chemotherapy regimen.
  Interventions: Drug: AB680; Drug: Nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: AB680 — AB680 is a Cluster of Differentiation (CD)73 Inhibitor.
Drug: Zimberelimab — Zimberelimab is a fully human immunoglobulin G4 (IgG4) monoclonal antibody targeting human PD-1.
  Other Names: AB122
  Arms: Dose Escalation; Dose Expansion (AB680 + zimberelimab + NP/Gem): Cohort B (second-line/2L); Dose Expansion (AB680 + zimberelimab + NP/Gem): Cohort C (front-line/1L); Dose Expansion (AB680+zimberelimab+ NP/Gem): Cohort A (front-line/1L); Dose Expansion (AB680+zimberelimab+NP/Gem):Cohort A1 (front-line/1L)
Drug: Nab-paclitaxel — Nab-paclitaxel is a chemotherapy agent. Chemotherapy agents are medicines that kill cancer cells.
  Other Names: Abraxane
Drug: Gemcitabine — Gemcitabine is a chemotherapy agent. Chemotherapy agents are medicines that kill cancer cells.
  Other Names: Gemzar

SUMMARY:
This is a Phase 1, open-label, dose-escalation, and dose-expansion, with a gated randomization portion, study to evaluate the safety, tolerability, pharmacokinetic, pharmacodynamic and clinical activity of AB680 in combination with zimberelimab (AB122), nab-paclitaxel and gemcitabine in participants with advanced pancreatic cancer.

DETAILED DESCRIPTION:
Dose escalation of AB680 in combination with zimberelimab (AB122), nab-paclitaxel and gemcitabine will be assessed in participants with advanced pancreatic cancer. In this dose escalation combination study, participants with advanced pancreatic cancer will receive escalating doses of AB680 in combination with zimberelimab at the recommended phase 2 dose (RP2D), and nab-paclitaxel and gemcitabine at standard doses. AB680, zimberelimab, nab-paclitaxel and gemcitabine are all administered via IV infusion.

In the dose expansion portion of the study in front-line (1L) pancreatic patients, participants will receive AB680 at the RP2D determined from the dose escalation study in combination with zimberelimab at the RP2D and nab-paclitaxel and gemcitabine at standard doses or AB680 at the RP2D in combination with nab-paclitaxel and gemcitabine at standard doses. In the dose-expansion portion of the study in second-line (2L) pancreatic patients, participants will receive AB680 at the RP2D determined from the dose-escalation study in combination with zimberelimab at the RP2D and nab-paclitaxel and gemcitabine at standard doses.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed metastatic pancreatic adenocarcinoma
* Naïve to any prior treatment, including chemotherapy, biological therapy, or targeted therapy for metastatic disease

  * Prior adjuvant therapy (including chemotherapy and/or radiotherapy) for pancreatic adenocarcinoma is permitted if neoadjuvant or adjuvant therapy was completed at least 6 months prior to study enrollment. Prior adjuvant therapy may include nab- paclitaxel or gemcitabine
  * Participants initially diagnosed with locally advanced pancreatic cancer who have undergone chemotherapy then resection and had no evidence of disease are eligible if relapse of metastatic disease has occurred and if the last dose of chemotherapy was received more than 6 months before study entry
* Must have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. The measurable lesion must be outside of a radiation field if the participant received prior radiation
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Confirmation that an archival tissue sample is available; if not, a new biopsy of a tumor must be obtained
* Prior radiation therapy for metastatic disease must have been completed
* Immunosuppressive doses of systemic medications, such as corticosteroids or absorbed topical corticosteroids (doses > 10 mg/day prednisone or equivalent) must be discontinued at least 2 weeks (14 days) before investigational product administration. Physiologic doses of corticosteroids (≤ 10 mg/day of prednisone or its equivalent) or short pulses of corticosteroids (≤ 3 days) may be permitted
* Prior surgery that required general anesthesia or other major surgery as defined by the Investigator must be completed at least 4 weeks before investigational product administration
* Negative tests for hepatitis B surface antigen, hepatitis C virus antibody (or hepatitis C qualitative ribonucleic acid [RNA; qualitative]), and human immunodeficiency virus (HIV)-1 and HIV-2 antibody at screening
* Adequate organ and marrow function

Key Exclusion Criteria:

* Significant cardiovascular disease (NYHA Class III-IV), myocardial infarction or cerebrovascular accident within 12 months of the first dose of investigational agent or history of arterial thromboembolic event, uncontrolled hypertension, unstable arrhythmia, or unstable angina within 3 months or venous thromboses within 1 month of the first dose of investigational agent.
* Any active autoimmune disease or a documented history of autoimmune disease or history of a syndrome that required systemic steroids or immunosuppressive medications, except for vitiligo or resolved childhood asthma/atopy. Participants with asthma who require intermittent use of bronchodilators (such as albuterol) will not be excluded from this study
* History of a syndrome that required systemic steroids or immunosuppressive medications, except for vitiligo or resolved childhood asthma/atopy. Participants with asthma who require intermittent use of bronchodilators (such as albuterol) will not be excluded from this study
* Prior malignancy active within the previous year except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix, breast, or prostate cancer
* Has not recovered (ie, ≤ Grade 1 or baseline) from a non-hematologic AEs due to a previously administered agent, except ≤ Grade 2 alopecia or ≤ Grade 2 neuropathy.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events (TEAEs) | From first dose date to 90 days after the last dose (approximately 1 year)
  Safety will be assessed by monitoring adverse events and clinically relevant changes in 12 lead Electrocardiogram (ECG) and Physical examination findings
Number of Participants With Dose Limiting Toxicities | From First dose to day 28

SECONDARY OUTCOMES:
Duration of response | Start date of response to first progression/death, up to 1 year
  Time at which response criteria are met for complete response or partial response (whichever occurs first) until the first date of recurrence, progression or death per RECIST v1.1
Disease control rate | First dose date to first progression/death
  Number of participants with complete response, partial response, or stable disease for greater than 6 months per RECIST v1.1
Overall survival | First dose date to date of death, up to 1 year
  Overall survival rate, defined as time between first dose date and date of death
Progression free survival | First dose date to first progression/death
  Number of participants without disease progression per RECIST v1.1
AB680 peak plasma concentration (Cmax) | Day 1 (sequential), day 2, day 3, day 8, day 15, day 29, day 36, day 43, day 57, day 85, day 197, day 309, day 421, 30 days after last dose, and 90 days after last dose
  Peak plasma concentration (Cmax) of AB680
Zimberelimab peak plasma concentration (Cmax) | Day 1 (sequential), day 2, day 3, day 8, day 15, day 29, day 43, day 57, day 85, day 197, day 309, day 421, 30 days after last dose, and 90 days after last dose
  Peak plasma concentration (Cmax) of zimberelimab
AB680 time of peak concentration (Tmax) | Day 1 (sequential), day 2, day 3, day 8, day 15, day 29, day 36, day 43, day 57, day 85, day 197, day 309, day 421, 30 days after last dose, and 90 days after last dose
  Time of peak concentration (Tmax) of AB680
Zimberelimab time of peak concentration (Tmax) | Day 1 (sequential), day 2, day 3, day 8, day 15, day 29, day 43, day 57, day 85, day 197, day 309, day 421, 30 days after last dose, and 90 days after last dose
  Time of peak concentration of zimberelimab
AB680 area under the plasma concentration versus time curve (AUC) | Day 1 (sequential), day 2, day 3, day 8, day 15, day 29, day 36, day 43, day 57, day 85, day 197, day 309, day 421, 30 days after last dose, and 90 days after last dose
  Area under the plasma concentration versus time curve (AUC) of AB680
Zimberelimab area under the plasma concentration versus time curve (AUC) | Day 1 (sequential), day 2, day 3, day 8, day 15, day 29, day 43, day 57, day 85, day 197, day 309, day 421, 30 days after last dose, and 90 days after last dose
  Area under the plasma concentration versus time curve (AUC) of zimberelimab
Immunogenicity indicators: anti-drug antibodies (ADA) | Day 1, day 15, day 29, day 57, day 85, day 197, day 309, and day 421
  Number of participants who develop anti-drug antibodies to zimberelimab
Overall response rate | First dose date to progression or last tumor assessment, up to 1 year
  Number of Participants with Complete or Partial Response per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v.1.1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences, Inc.
Locations (17):
- United States (17):
  - The Angeles Clinic, Los Angeles, California
  - UCLA Hematology Oncology, Santa Monica, California
  - Yale Cancer Center, New Haven, Connecticut
  - BRCR Global, Plantation, Florida
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - NYU Cancer Institute, New York, New York
  - Columbia University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Canon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - START San Antonio, San Antonio, Texas
  - Medical Oncology Associates, Spokane, Washington
  - UW Health - UW Carbone Cancer Center - Medical Oncology Clinic, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- See also: ARC-8 - Public website — https://trials.arcusbio.com/study/?id=ARC-8